CLINICAL TRIAL: NCT05487989
Title: Study of the VIsual Pathways MODEL for a Better Understanding of Neurodegeneration in Inflammatory and Demyelinating Disorders of Central Nervous System
Brief Title: VIsual Pathways Model in Neuro-inflammatory Disorders
Acronym: VIP-MODEL
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0289; 2022-A01483-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-07-11; First posted 2022-08-04 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Optic Neuritis
Keywords: Optic neuritis; Optical coherence tomography, MRI, demyelination, neuro-axonal loss.; MRI; demyelination; neuro-axonal loss
MeSH Terms: conditions — Optic Neuritis; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- optic neuritis patients: Patients suffering from an acute episode of optic neuritis will be included. There will be only one group of patients prospectively followed-up.
  Interventions: Other: Clinical examen

INTERVENTIONS:
Other: Clinical examen — MRI sequences for research, pupillometry, OCT-angiography, evaluation of visual cognition

SUMMARY:
In neuroinflammatory diseases of the central nervous system (CNS) such as multiple sclerosis (MS), neuromyelitis optica spectrum disorders (NMOSD) and anti-MOG antibody-associated disorders (MOGAD), neuronal degeneration is the consequence of inflammatory and demyelinating lesions in the brain, optic nerve and spinal cord. Both white and grey matter are systematically affected. Lesions of the perivascular spaces containing cerebrospinal fluid (CSF) and meningeal inflammation seem to play an important role in the pathophysiology of these neuroinflammatory diseases. Currently, the interrelation of all these aspects is not clearly established in the pathophysiology of these diseases. In order to better understand the mechanisms that lead to and underlie the clinical disability of patients with these diseases, we need in vivo study models that allow the in-depth study of the neurodegenerative process and the identification of its causes. In this perspective, we make the hypothesis that the visual pathways model is very relevant to measure neuro-axonal loss and to explore the different mechanisms involved in neurodegeneration during MS and other CNS demyelinating diseases. Researchers have at their disposal many tools that allow them to analyse and quantify the neurodegenerative process in a reproducible and very precise manner from a structural and functional point of view, while taking into account possible vascular involvement (MRI, optical coherence tomography - angiography, etc…).

ELIGIBILITY:
Inclusion Criteria:

* - Male or female
* Aged between 18 and 65 years
* Presenting a clinical picture of optic neuritis for less than 4 weeks, confirmed by neuro-ophthalmological assessment
* Patient having given written consent to participate in the study
* Patient with social insurance
* Patient willing to comply with all study procedures and duration

Exclusion Criteria:

* - history of optic neuritis on the same side as the recent episode for which the patient is being treated
* history of retinal pathology (retinal detachment, glaucoma, retinopathies, retinal surgery)
* diabetes
* chronic alcohol intoxication
* contraindications to MRI
* pregnant women
* persons under protective supervision (ex : guardianship)
* minors
* persons deprived of their liberty
* administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of social security coverage, refusal to sign consent

A history of pre-existing CNS inflammatory demyelinating disease is not a criterion for non-inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting an episode of acute optic neuritis with the objective of better understanding the pathophysiology of CNS inflammatory diseases and identifying prognostic biomarkers in imaging
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2028-04-07 (Estimated)

PRIMARY OUTCOMES:
Presence of enhancement of the optic nerve sheath on the axial T1 dixon MRI sequence post gadolinium at the acute phase of optic neuritis. | at inclusion
Low contrast monocular visual acuity (2.5%, LogMAR unit) at distance from acute optic neuritis | at 12 months

SECONDARY OUTCOMES:
Presence of enhancement of the optic nerve sheath on the axial T1 dixon MRI sequence post gadolinium. Macular GCIPL atrophy will be assessed by the variation of mGCIPL volume between inclusion and the maximal follow-up. | at inclusion and at 12 months follow-up
Optic nerve lesion length on 3D-DIR sequence. Alteration of retinal microvascularisation between inclusion and the maximal follow-up. | at inclusion and at 12 months follow-up
Acute alteration of retinal microvascularisation is assessed by the difference of retinal vascular density between inclusion (V0) and one month later (V1). | at inclusion and at 1 months follow-up
Low contrast monocular visual acuity (2.5%, LogMAR unit) measured at 12 months (V5) | at inclusion and at 12 months follow-up
Amplitude of the melanopsin-mediated sustained constriction phase in the blue light-induced pupillary response is assessed at 12 months (V5). | at inclusion and at 12 months follow-up
Optic nerve lesion length assessed at inclusion (V0) | at inclusion
mGCIPL atrophy/retinal vascular alteration are assessed by mGCIPL volume/retinal vessel density difference between inclusion (V0) and at 12 months (V5). | at inclusion and at 12 months follow-up
Presence of leptomeningeal cerebral enhancement | at inclusion, at 6 months and at 12 months follow-up
T2 lesions brain and spinal cord volumes | at inclusion, at 6 months and at 12 months follow-up
Brain grey matter volumes and brain perfusion (3D-ASL) | at inclusion, at 6 months and at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Olivier OUTTERYCK, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Fontan Chu, Lille, France